CLINICAL TRIAL: NCT02379234
Title: SIMulation for HEmofiltration in Intensive caRe Unit
Brief Title: Simulation for Continuous Veno-venous Hemofiltration in Intensive caRe
Acronym: SIMHeR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 49RC13_0209
Record Dates: First submitted 2015-02-12; First posted 2015-03-04 (Estimated); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Hemofiltration; Nurse Training; Health Care Provider Education
Keywords: CVVH; Renal replacement therapy; High fidelity simulation; Nurse training

STUDY DESIGN:
Intervention Model Description: We performed a 2-phase (training and evaluation), randomized, single-center, open study: During the training phase, intensive care unit nurses underwent a 6-hour training pro- gram and were randomized to receive (intervention) or not (control) an additional high-fidelity simulation training (6 hours). During the evaluation phase, management of CRRT sessions was randomized to either intervention or control nurses.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): All nurses received a 4 hours formation, called "conventional formation", given by a professional trainer, that included 2 hours of theorical formation and 2 hours of practical training, based on CVVH generator demonstration. In addition, the trainer was present in the ICU during the first week of CVVH implementation, to answer any questions and to help nurses with their first CVVH sessions
- Simulated (Experimental): The 'Simulated formation',used high fidelity mannequin and CVVH generator, is composed of 3 training sessions of 2 hours each one. This formation is associated with the 'conventional formation'.
  Interventions: Other: simulation

INTERVENTIONS:
Other: simulation — Nurses received, in addition to the conventional formation (as in the control arm), a set of 3 high-fidelity simulation sessions. Each session lasted 1 to 2 hours, used high fidelity mannequin and CVVH generator and took place in an ICU room environment. For each session, a specific scenario was designed, the session began with a briefing and ended with a debriefing, based on video recording.
  Arms: Simulated

SUMMARY:
Continuous Veno-Veinous Hemofiltration (CVVH) is a frequently used renal replacement therapy in intensive care units for patients with acute renal failure. In theory, this therapy should be continuous, 24 hours/day.

However, it is wellknown that actual duration of CVVH sessions is much lower than scheduled, with frequent "circuit down-times" (between 1 to 6 hours/day). There are many reasons for premature ending of CVVH sessions (i.e. catheter dysfunction, wrong settings, low anticoagulation…), but early detection of any dysfunction may prevent (at least in part) the CVVH circuit coagulation. ICU Nurses are on the first line to manage CVVH sessions, particularly in case of alarms.

High-fidelity simulation has been recently proposed for health care provider education. It has been consistently associated with large effects for outcomes of knowledge, skills, and behaviors but with moderate effects for patient related outcomes. Indeed, few studies have assess the impact of simulation on patient outcome following complexe procedures, that implies team work in addition to individual skills.

In our 12-bed surgical ICU, investigators have decided to implement CVVH technics (in addition to the dialysis that we already used). Before implementing this new technic in the ICU, investigators designed this study in order assess wether a high-fidelity based ICU-nurses education program would improve the outcome of CVVH sessions, compared to the conventional education program, proposed by the CVVH manufacturer.

DETAILED DESCRIPTION:
All nurses of our 12-beds surgical ICU were randomized to one of the two arms for CVVH training (ie "conventional", the control arm, or "conventional + high-fidelity simulation", the intervention arm). Randomization was stratified according to nurse's experience with dialysis (i.e. defined as novice, standard or expert).

Then, all CVVH sessions performed in the ICU, were randomized to be supervised by nurses of one of the two arms only. The nurse in charge of the patient could thus be changed, depending on his/her group (note that the usual ratio is 1 nurse for 2.5 patients). Investigators use a minimization algorithm for this randomization, that take into account the presence of shock, counter-indication for heparin use, patient's agitation, site of dialysis catheter insertion (ie. Internal jugular or femoral) and previous early ending of the session. Prescription of CVVH was standardized (ie. Objective of 35 ml/kg/h of ultrafiltrate, with 1/3 in predilution and 2/3 post-dilution), and used unfractionated heparin.

All CVVH parameters (i.e. pressures, flow, alarms…) were recorded continuously, using a computer. In addition, hemodynamic parameters and biological parameters were prospectively recorded every 3 hours.

Prescription of CVVH ending should be timely written by the doctors. Nurses were asked to clearly record the time of CVVH session ending. An ending appearing less than 4 hours before the scheduled arrest of the session is considered as a "prematurely ending". Total and effective duration of each session were also recorded , as well as the total volume of ultrafiltrate.

ELIGIBILITY:
Inclusion Criteria:

- All ICU-nurses were recruited.

Exclusion criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2014-01; Primary Completion 2016-09-01 (Actual); Study Completion 2016-09-01 (Actual)

PRIMARY OUTCOMES:
percentage of CVVH sessions ended prematurely as measured by a percentage | Two years

SECONDARY OUTCOMES:
Management of CVVH generator alarms during the sessions as measured by the number of 'calling for help' during the session | 72 hours
efficacy of CVVH session measured by creatinine and bilirubin rate | 72 hours
Evaluation of nurses satisfaction measured by a quiz | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Sigismond Lasocki, Principal Investigator — University Hospital, Angers
Locations (1):
- Pr Lasocki Sigismond, Angers, France

REFERENCES:
- [Result] Lemarie P, Husser Vidal S, Gergaud S, Verger X, Rineau E, Berton J, Parot-Schinkel E, Hamel JF, Lasocki S. High-Fidelity Simulation Nurse Training Reduces Unplanned Interruption of Continuous Renal Replacement Therapy Sessions in Critically Ill Patients: The SimHeR Randomized Controlled Trial. Anesth Analg. 2019 Jul;129(1):121-128. doi: 10.1213/ANE.0000000000003581. PMID 29933269